CLINICAL TRIAL: NCT03564704
Title: An Open-Label, One-Arm, Multi-Site Trial of Precision Diagnosis Directing Histone Deacetylase Inhibitor Chidamide Total Therapy for Adult T-lymphoblastic Lymphoma/Leukemia
Brief Title: Precision Diagnosis Directing HDACi Chidamide Target Therapy for Adult T-LBL/ALL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, M.D., Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDT-ALL-LBL
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Leukemia; Leukemia, Acute; Adult Lymphoblastic Lymphoma; Leukemia, Lymphoblastic; Leukemia, T Cell; Adult Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma; Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, T-Cell | interventions — Dexamethasone; Vincristine; Cyclophosphamide; Idarubicin; pegaspargase; Doxorubicin; Methotrexate; Mercaptopurine; Etoposide; Cytarabine; Injections, Spinal; Radiotherapy; Karyotyping; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PDT-ALL-LBL (Experimental): The intervention of PDT-ALL-LBL consists of diagnostic test (bone marrow aspiration, flow immunophenotyping, karyotyping，FISH, NGS, Flow-MRD, PET-CT scan), induction regimen (chidamide, dexamethasone, vincristine, cyclophosphamide, idarubicin, pegaspargase), consolidation regimen (chidamide, prednisone, cytarabine, methotrexate, cyclophosphamide, etoposide, adriamycin, 6-mercaptopurine, pegaspargase), MRD assessment and maintenance regimen (chidamide, prednisone, vincristine, methotrexate, 6-mercaptopurine), intrathecal injection chemotherapy (methotrexate, cytarabine, dexamethasone), radiation therapy (for mediastinum- and/or central nervous system-involved lymphoma/leukemia) and allogeneic hematopoietic stem cell transplantation for patients with donor.
  Interventions: Drug: Dexamethasone; Drug: vincristine; Drug: Cyclophosphamide; Drug: Idarubicin; Drug: Pegaspargase; Drug: Adriamycin; Drug: Methotrexate; Drug: 6-mercaptopurine.; Drug: Etoposide; Drug: Cytarabine; Procedure: Bone marrow aspiration; Procedure: Intrathecal injection; Radiation: Radiation therapy; Genetic: NGS; Procedure: allogeneic hematopoietic stem cell transplantation; Diagnostic Test: Flow-MRD; Diagnostic Test: FISH; Diagnostic Test: Flow immunophenotyping; Diagnostic Test: Karyotyping; Drug: Chidamide; Diagnostic Test: PET-CT scan

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone will be added in Pre-phase Regimen, Induction-Regimen, Consolidation-Module of PDT-ALL-LBL protocol.
  Other Names: DXM
Drug: vincristine — Vincristine will be added to Induction-Regimen, Consolidation-Module and Maintenance-Module of PDT-ALL-LBL protocol.
  Other Names: VCR
Drug: Cyclophosphamide — CTX will be added to Induction-Regimen, Consolidation-Module and Maintenance-Module of PDT-ALL-LBL protocol.
  Other Names: CTX
Drug: Idarubicin — IDA will be added to Induction-Regimen and Consolidation-Module of PDT-ALL-LBL protocol.
  Other Names: IDA
Drug: Pegaspargase — PEG-ASP will be added to Induction-Regimen and Consolidation-Module of PDT-ALL-LBL protocol.
  Other Names: PEG-ASP
Drug: Adriamycin — Adriamycin will be added to Consolidation-Module of PDT-ALL-LBL protocol.
  Other Names: ADR
Drug: Methotrexate — Methotrexate will be added to Consolidation-Module of PDT-ALL-LBL protocol.
  Other Names: MTX
Drug: 6-mercaptopurine. — Mercaptopurine will be added to Consolidation-Module and Maintenance-Module of PDT-ALL-LBL protocol.
  Other Names: 6-MP
Drug: Etoposide — VP-16 will be added to Consolidation-Module of PDT-ALL-LBL protocol.
  Other Names: VP-16
Drug: Cytarabine — AraC will be added to Consolidation-Module of PDT-ALL-LBL protocol.
  Other Names: AraC
Procedure: Bone marrow aspiration — Bone marrow aspiration and additional tests will be performed in all module of PDT-ALL-LBL protocol.
  Other Names: BM smear
Procedure: Intrathecal injection — Intrathecal injection of chemotherapy will be performed in PDT-ALL-LBL protocol.
  Other Names: IT
Radiation: Radiation therapy — Radiation therapy will be performed for mediastinum and/or central nervous system leukemia/lymphoma in PDT-ALL-LBL protocol.
  Other Names: RT
Genetic: NGS — Next-Generation-Sequencing (NGS) will be performed in PDT-ALL-LBL protocol.
Procedure: allogeneic hematopoietic stem cell transplantation — Allo-HSCT will be added to LBL patients with available donor in PDT-ALL-LBL protocol.
  Other Names: Allo-HSCT
Diagnostic Test: Flow-MRD — Flow-MRD will be added to PDT-ALL-LBL for bone marrow and cerebrospinal fluid samples.
Diagnostic Test: FISH — FISH will be added to PDT-ALL-LBL for bone marrow samples.
Diagnostic Test: Flow immunophenotyping — Flow immunophenotyping will be performed in PDT-ALL-LBL protocol.
Diagnostic Test: Karyotyping — Karyotyping will be performed in PDT-ALL-LBL protocol.
Drug: Chidamide — HDACi chidamide will be added to induction regimen, consolidation and maintenance module of PDT-ALL-LBL.
  Other Names: HDACi Chidamide
Diagnostic Test: PET-CT scan — PET-scan will be performed for T-LBL patients for MRD assessment in PDT-ALL-LBL.
  Other Names: PET-CT

SUMMARY:
Based on the pediatric-inspired, PEG-L-asparaginase-intensified and MRD-directed PDT-ALL-2016 protocol, this open-label, one-arm, multi-site trial PDT-ALL-LBL is aimed to evaluate the safety and effect of oral histone deacetylase inhibitor chidamide for adult T-ALL/LBL. Compared to PDT-ALL-2016 for B-ALL, HDACi chidamide will be administrated from induction therapy to maintenance therapy, along with higher dose of consolidation regimen of cytarabine, methotrexate, cyclophosphamide.

DETAILED DESCRIPTION:
T-lymphoblastic lymphoma/leukemia is a neoplasm of lymphoblasts committed to the T-cell lineage, typically composed of small to medium-sized blast with scant cytoplasm, moderately condensed to dispersed chromatin, and inconspicuous nucleoli, involving bone marrow and blood or presenting with primary involvement of the thymus or of nodal or extranodal sites. T-ALL/LBL is generally considered a higher-risk disease than B-ALL. Compared to B-ALL, T-LBL/ALL is associated with a higher risk of induction failure, early relapse, and isolated CNS relapse.

Chidamide is a novel oral HDACi with promising activity in non-Hodgkin lymphoma (NHL). Chidamide, a new oral isotype-selective HDACi, approved in China for the treatment of R/R PTCL in December 2014. Based on the pediatric-inspired, PEG-L-asparaginase-intensified and MRD-directed PDT-ALL-2016 protocol, this open-label, two-arm, multi-site trial PDT-ALL-LBL is aimed to evaluate the safety and effect of oral histone deacetylase inhibitor chidamide for adult T-ALL/LBL. Compared to PDT-ALL-2016 for B-ALL, HDACi chidamide will be administrated from induction therapy to maintenance therapy, along with higher dose of consolidation regimen of cytarabine, methotrexate, cyclophosphamide.

The intervention of PDT-ALL-LBL consists of diagnostic test (bone marrow aspiration, flow immunophenotyping, karyotyping，FISH, NGS, Flow-MRD), induction regimen (chidamide, dexamethasone, vincristine, cyclophosphamide, Idarubicin, pegaspargase), consolidation regimen (chidamide, prednisone, cytarabine, methotrexate, cyclophosphamide, etoposide, adriamycin, 6-mercaptopurine, pegaspargase), MRD assessment (MRD1/d14, MRD2/d24, MRD3/d45, MRD4/pre-allo-HSCT) and maintenance regimen (chidamide, vincristine, methotrexate, 6-mercaptopurine), intrathecal injection, radiation therapy (for mediastinum- and/or central nervous system-involved lymphoma/leukemia) and allogeneic hematopoietic stem cell transplantation for patients with donor.

Induction Regimen-Pretreatment: dexamethasone, -3d to 0d; Induction regimen VICLD: VCR: d1, d8, d15, d22; IDA: d1, d8; CTX: 1g/m2, 1; PEG-asp: 2000-2500IU/m2, 1, 15; dexamethasone: 1-24; chidamide: 10mg/d, po, qd. Flow-based MRD assessment: d14, d24 during induction regimen, d45, and pre-HSCT. Salvage regimen VLCAM (MRD1/d24>1%): CTX, d25; AraC 50mg/m2, d25-31; 6-MP: 25-31, PEG-asp: 2500IU/m2, d26. Consolidation Module (CM)-CM1: AraC 3g/m2, q12h, d1-2, Dex: 10mg/m2, d1-2, PEG-asp: 2, 6-MP: d1-7, chidamide, po qd; CM2: MTX 5g/m2, 1, Dex: 10mg/m2, 1-2, PEG-asp: d2, 6-MP: 1-7, chidamide, po qd; CM3: CTX 1g/m2, 1-3, PEG-asp: 2, 6-MP: 1-7, chidamide, po qd. CM4-6: repeat CM 1-3. Re-Induction: VICLD after CM6. CM7-9: repeat CM1-3. Allo-HSCT: after CM3 when matched-related-donor (MRD), haploidentical related donor (HRD) or matched-unrelated-donor (MUD) available. Non-allo-HSCT: finish CM4-9 and CPOMP maintenance. Maintenance Module-CPOMP: chidamide, po qd for 24 months; Pred: for 12 months; VCR for 12 months; MTX: for 24m months; 6-MP for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* 14-55 years old;
* LBL/ALL newly diagnosed;
* signed written informed consent.

Exclusion Criteria:

* Pregnant women;
* History of pancreatitis;
* History of diabetes;
* History of active peptic ulcer disease in the past 6 months;
* History of arteriovenous thrombosis in the past 6 months;
* Severe active infection;
* Allergic to any drugs in PDT-ALL-LBL protocol.

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-02-14 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Event-Free-Survival | 3 years
  3 years EFS of LBL/ALL patients enrolled in PDT-ALL-LBL

SECONDARY OUTCOMES:
Minimum residual disease after induction | 3 months
  MRD after induction regimen of PDT-ALL-LBL protocol
CR after Induction Therapy | 3 months
  CR after induction regimen of PDT-ALL-LBL protocol
Death in induction | 3 months
  Dearth during induction regimen of PDT-ALL-LBL
Adverse events | 3 years
  AE of 3 years of LBL patients enrolled in PDT-ALL-LBL
Relapse | 3 years
  Cumulative incidence relapse rate of 3 years of LBL patients enrolled in PDT-ALL-LBL protocol
Relapse free survival | 3 years
  3 years RFS of LBL patients enrolled in PDT-ALL-LBL protocol
Overall survival | 3 years
  3 years OS of LBL patients enrolled in PDT-ALL-LBL protocol

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD, Study Chair — Department of Hematology Nanfang Hospital
Locations (1):
- Department of Hematology, Nanfang Hospital, Guangzhou, Guangdong, China